CLINICAL TRIAL: NCT04452942
Title: Dynamic Changes in Cytokine and Eicosanoid Mediators Among Hospitalized Patients With Coronavirus Infectious Disease 2019 (COVID-19)
Brief Title: Cytokine and Eicosanoid Mediators in Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: EicOsis Human Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EC1153-2-01
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Coronavirus Disease 2019; SARS-CoV-2; Eicosanoids; Eicosanoid storm; Cytokine storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, single center, observational, cohort study of patients to (1) describe the kinetics and temporal relationship of changes in eicosanoid and cytokine mediators in patients with severe COVID-19 admitted to the hospital; and (2) correlate the dynamic changes in eicosanoid mediators with available patient clinical status, including measures of severity of illness, routine laboratory tests, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with symptoms suggestive of COVID-19.
2. Confirmed infection with SARS-CoV-2 as determined by polymerase chain reaction (PCR) or other commercial or public health assay in the 72 hours prior to hospital admission or any time during hospital admission.
3. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
4. Understands and agrees to comply with planned study procedures.
5. Agrees to the collection of whole blood samples.

Exclusion Criteria:

1. Inability to obtain informed consent.
2. Anticipated transfer to another hospital which is not a study site within 48 hours.
3. Inability to obtain sequential blood samples due to patient's characteristics (i.e. difficult vascular access).
4. Obstetric patients.
5. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with laboratory-confirmed SARS-CoV-2 infection requiring hospitalization for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Changes on eicosanoid lipid mediators | 10 days
  Temporal changes on eicosanoid lipid mediators over a course of 10 days (or until discharge) in COVID-19 patients requiring hospitalization
Changes on plasma levels of a panel of 40 human cytokines and chemokines | 10 days
  Temporal changes on the levels of 40 human cytokines, chemokines and growth factors included in a commercially available panel (Bio-Rad, Human Chemokine Panel, 40-Plex #171AK99MR2) over a course of 10 days (or until discharge) in COVID-19 patients requiring hospitalization.

SECONDARY OUTCOMES:
Severe clinical outcome | Through study completion, an average of 10 days
  Severe clinical outcome defined as need for ICU admission and/or need for mechanical ventilation and/or multi-organ failure and/or death during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.eicosis.com